CLINICAL TRIAL: NCT00973284
Title: Phase 1-2, Randomized, Multi-Center, Double-Blind, Placebo-Controlled, Safety and Efficacy Study in Healthy Adults of Intranasal Norwalk Virus-like Particle Vaccine in Experimental Human Norwalk Virus Infection
Brief Title: Norwalk Vaccine Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LV01-103; U1111-1176-0535 (Registry Identifier: WHO)
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Acute Gastroenteritis; Norwalk Virus Infection
Keywords: Prevention of acute gastroenteritis due to infection with and experimental Norwalk Virus
MeSH Terms: interventions — Mannitol; Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Norwalk VLP Vaccine 100 µg (Experimental): Norwalk Virus-like Particle (VLP) Vaccine 100 µg, dry powder, intranasally using a delivery device with a puff of air, 50 µg in each nostril, on Days 0 and 21 in the Vaccination Stage. Norwalk Virus, 48 Reverse Transcription Polymerase Chain Reaction (RT-PCR) units, solution, orally, on Day 42 in the Challenge Stage.
  Interventions: Biological: Norwalk VLP vaccine; Biological: Norwalk virus
- Placebo (Placebo Comparator): Norwalk VLP placebo-matching vaccine, dry powder, intranasally using a delivery device with a puff of air, 50 µg in each nostril, on Days 0 and 21 in the Vaccination Stage. Norwalk Virus, 48 RT-PCR units, solution, orally, on Day 42 in the Challenge Stage.
  Interventions: Biological: mannitol and sucrose; Biological: Norwalk virus

INTERVENTIONS:
Biological: Norwalk VLP vaccine — Norwalk VLP vaccine dry powder
  Arms: Norwalk VLP Vaccine 100 µg
Biological: mannitol and sucrose — Mannitol and sucrose as placebo-matching Norwalk VLP Vaccine dry powder
  Arms: Placebo
Biological: Norwalk virus — Norwalk virus solution

SUMMARY:
The purpose of this study was to evaluate the efficacy of the Norwalk virus-like particle (VLP) vaccine as determined by the illness rate of viral acute gastroenteritis (AGE) during the inpatient stay.

DETAILED DESCRIPTION:
The drug being tested in this study is called intranasal Norwalk virus-like particle (VLP) vaccine. Norwalk VLP vaccine is being tested to prevent viral acute gastroenteritis (AGE). This study will look at the illness rate of AGE in people who are administered the Norwalk VLP vaccine.

The study enrolled 98 patients and was conducted in 2 stages: the Vaccination Stage and the Challenge Stage. In the Vaccination Stage participants were randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which remained undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Norwalk VLP Vaccine (100 µg VLP) intranasally
* Placebo (dummy inactive powder) - this is a powder that looks like the study drug but has no active ingredient During the Challenge Stage participants were administered live Norwalk virus and were monitored for AGE.

This multi-center trial was conducted in the United States. The overall time to participate in this study was up to 29 weeks Participants made multiple visits to the clinic and were contacted by telephone 6 months after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consents.
2. Age 18 - 50 years, inclusive.
3. Good general health as determined by a screening evaluation within 45 days of randomization.
4. Expressed interest, availability, and understanding to fulfill the study requirements including measures to prevent Norwalk virus contamination of the environment and spread of infection and illness to the community. The prospective subjects must pass (> 75 % correct answers) a written examination on all aspects of the study before enrollment. (Appendix D)
5. Available to return for follow-up visits following discharge from the inpatient unit and deliver stool specimens to the investigator promptly.
6. Female subjects must be of non-childbearing potential, or if of childbearing potential (as determined by the investigator) must be practicing abstinence or using an effective licensed method of birth control (e.g. oral contraceptives; diaphragm or condom in combination with contraceptive jelly, cream, or foam; intrauterine contraceptive device, or Depo-Provera; skin patch; vaginal ring or cervical cap) for 30 days prior to vaccination and must agree to continue such precautions during the study and for 60 days after the Challenge visit. Male subjects must agree not to father a child during the study and for 60 days after the Challenge visit.
7. Demonstrated to be H type-1 antigen secretor positive (by saliva test). [This saliva test may be done outside of the 45 day window and does not need to be repeated.]
8. Agrees not to participate in another clinical trial with an investigational product for the entire duration of the study (six months after the last dose of study vaccine or placebo i.e. 201 days).

Exclusion Criteria:

1. Living with or having daily contact with children age 5 years or less or a woman known to be pregnant. This includes significant contact at home, school, day-care, or equivalent facilities.
2. Nursing mother.
3. Living with or having daily contact with childcare workers.
4. Living with or having daily contact with elderly persons aged 70 years or more, or infirmed, diapered individuals, persons with disabilities or incontinent persons. This includes work or visits to nursing homes and day-care or equivalent facilities.
5. Evidence of recent (within 2 months) or of current nonbacterial gastroenteritis suggestive of Norwalk virus infection [vomiting or unformed or watery stools ( > 2 during a 24 hour period)].
6. Any gastroenteritis within the past 2 weeks.
7. History of chronic functional dyspepsia, chronic gastroesophageal reflux disease, peptic ulcer disease, gastrointestinal hemorrhage, gall bladder disease, inflammatory bowel disease, irritable bowel syndrome, frequent diarrhea, chronic constipation, or diverticulitis anytime during the subject's lifetime.
8. Regular use of medication other than oral contraceptive agents, anti-hypertensives, anti-depressants, vitamins and minerals.
9. History of any of the following medical illnesses:

   * Chronic rhinitis, runny nose, sneezing (including seasonal allergies)
   * Clinically significant nose bleed within the prior 12 months
   * Diabetes
   * Cancer (malignancies other than a resolved skin lesion)
   * Heart disease (hospitalization for a heart attack, arrhythmia, or syncope)
   * Unconsciousness (other than a single brief "concussion")
   * Seizures (other than febrile seizures as a child <5 years old)
   * Asthma requiring treatment with inhaler or medication in the prior 2 years
   * Neuro-inflammatory disease
   * Autoimmune disease
   * Eating disorder
   * Chronic headaches associated with vomiting
   * Chronic vomiting syndrome
10. Any current illness requiring daily medication other than vitamins, minerals, birth control, anti-depressants or anti-hypertensives.
11. Blood Type B or AB. [This blood test may be done outside of the 45 day window and does not need to be repeated.]
12. Allergies or hypersensitivity to chitosan, shrimp, other shellfish or any component of the vaccine or placebo.
13. History of nasal surgery of any type (including tonsillectomy or adenoidectomy).
14. Any clinically significant abnormality detected on physical examination, including:

    * Murmur (other than a functional murmur)
    * Focal neurological abnormality
    * Hepatosplenomegaly
    * Lymphadenopathy
    * Jaundice
15. Hypertension defined as BP > 150/90 mm Hg on two separate measurements. Chronic stable well-controlled hypertension on medications is allowed.
16. History of more than 3 hospitalizations for invasive bacterial infections (pneumonia, meningitis), acute or chronic dermatitis (e.g. eczema, seborrhea, psoriasis) or collagen vascular disease [e.g. systemic lupus erythematosus (SLE) or dermatomyositis].
17. Presence of other serious chronic illness (i.e. malignancy other than a resolved skin lesion).
18. Positive stool/fecal culture for bacterial pathogens (salmonella, campylobacter, E. coli 0157:H7, and shigella) or positive stool/fecal screen for ova and parasites.
19. Employment in the food service industry, such as restaurants, or cafeteria facilities. Specifically, this will include persons whose employment requires food processing in the 4 weeks following challenge.
20. Health-care workers with patient contact expected in the 4 weeks following challenge.
21. Expected contact (through employment or at home) with immunocompromised persons (HIV-positive, receiving immunosuppressive medications such as oral steroids, anti-neoplastic agents) in the 4 weeks following challenge.
22. Employment as an airline flight attendant, scheduled to work in the 4 weeks following challenge.
23. Persons planning on taking a cruise in the 4 weeks following challenge.
24. Persons who have consumed or plan to consume raw shellfish (e.g. oysters) within 7 days prior to enrollment or throughout the study.
25. Any of the following lab abnormalities:

    * Absolute neutrophil count (ANC) or total white blood cell (WBC) outside the normal range (may be repeated once if outside this limit)
    * Hemoglobin outside the normal range (may be repeated once if outside this limit)
    * Platelet count outside the normal range (may be repeated once if outside this limit)
    * Electrolytes, blood urea nitrogen (BUN) and/or creatinine outside the normal range (may be repeated once if outside this limit)
    * Glucose > upper limit of normal (ULN) (may be repeated once if outside this limit). Fasting glucose is not required.
    * Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, bilirubin (total and indirect) or gamma glutamyl transferase (GGT) outside the normal range (may be repeated once if outside this limit)
    * Positive serology for hepatitis C or human immunodeficiency virus (HIV) antibody or hepatitis B surface antigen or rapid plasma reagin (RPR)
26. For women, positive serum pregnancy test within 14 days or positive urine pregnancy test within 24 hours of randomization.
27. Temperature > 99.7°F orally or symptoms of an acute self-limited illness such as an upper respiratory infection or gastroenteritis within 3 days of randomization.
28. Previous participation in a study of experimental norovirus infection or vaccines.
29. Study site personnel or their family members.
30. Significant history of psychiatric hospitalization, alcohol abuse, or illicit drug use.
31. Receipt of a licensed live vaccine within 28 days or a licensed inactivated vaccine within 14 days of randomization.
32. Completion of an investigational vaccine or drug study within 28 days of randomization.
33. Other condition that in the clinical judgment of the investigator would jeopardize the safety or rights of a subject participating in the trial, would render the subject unable to comply with the protocol or would interfere with the evaluation of the vaccination stage or the evaluation of the challenge stage.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2009-08-04 (Actual); Primary Completion 2010-04-07 (Actual); Study Completion 2010-08-18 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Viral Acute Gastroenteritis (AGE) | 7 Days Post-Challenge
  Viral AGE was a composite endpoint for the analysis of clinical illness and was defined as meeting one or more definitions of Norwalk Virus Infection and one or more of the definitions of AGE.
  Norwalk Virus Infection:
  * PAN-Immunoglobulin (Ig) Enzyme Linked Immunosorbent Assay (ELISA) for anti-Norwalk Virus Antibody IgM, IgG and IgA, ≥4-fold rise in titer in serum on Challenge Day 30 compared to Pre-Challenge.
  * Reverse Transcription Polymerase Chain Reaction (RT-PCR), a single positive post-challenge stool sample.
  * Norwalk Virus Antigen, a single positive post-challenge stool sample.
  Acute Gastroenteritis:
  ->200 grams of watery feces in 24-hour collection that immediately takes the shape of the container.
  * Vomiting and watery feces ≤200 grams on the same or consecutive days.
  * One vomiting episode plus one of the following symptoms: abdominal cramps or pains, nausea, bloating, loose feces, fever ≥99.7° Fahrenheit, or myalgia on the same or consecutive days.

SECONDARY OUTCOMES:
Percentage of Participants with Norwalk Virus Infection Anytime Post Challenge | Up to 30 Days Post-Challenge
  Norwalk Virus Infection was defined as meeting one or more of the following criteria:
  * Norwalk Virus Antigen, a single positive post-challenge stool sample.
  * Reverse Transcription Polymerase Chain Reaction (RT-PCR), a single positive post-challenge stool sample.
  * PAN-Immunoglobulin (Ig) Enzyme Linked Immunosorbent Assay (ELISA) for anti-Norwalk Virus Antibody IgM, IgG and IgA, ≥4-fold rise in titer in serum on Challenge Day 30 compared to Pre-Challenge.
Severity of Viral AGE using the Modified Vesikari Scale | Up to 30 Days Post-Challenge
  Vesikari Scoring System assesses the following symptoms: duration of diarrhea (days), maximum number of diarrheal stools/24 hours, duration of vomiting (days), maximum number of vomiting episodes/24 hours, fever and dehydration. Since the typical inpatient phase was four days in length, the duration of diarrhea scoring was modified to fit this time frame. Modified Vesikari Scale Total Score=17. Higher numbers are worse.
Duration of Viral AGE Among Challenged Participants | Up to 30 Days Post-Challenge
  Duration of symptoms was determined by a blinded committee review of each participant's symptoms. Participants not ill are included in the calculations with a duration=0.
Percentage of Participants with Norwalk Virus Antigen Detected in the Stool | Days 1 thru 4, 7, 21 and 30 in the Challenge Stage
  Stool samples were collected following challenge with Norwalk Virus. A positive test for antigen in post challenge stool sample was considered evidence of Norwalk Virus infection.
Percentage of Participants with Seroconversion in Serum Anti-Norwalk Virus | Pre-Challenge to 30 Days Post-Challenge
  Seroconversion was defined as a 4-fold rise in Pan-Ig ELISA Assay (Combined IgG + IgA + IgM) from Pre-Challenge to Day 30 Post Challenge.
Percentage of Participants with Norwalk RT-PCR Positive Titer in Stool Anytime Post Challenge | Days 1 thru 4, 7, 21 and 30 in the Challenge Stage
  RT-PCR was carried out to detect Norwalk Virus RNA in stool samples. A single positive test was taken as evidence of a Norwalk Virus infection.
Percentage of Participants with Any Local Intranasal Symptoms during the Vaccination Stage | 7 Days Post Dose 1 and 2
  Local symptoms included nasal stuffiness, nasal itching, sneezing, runny nose/nasal discharge, nasal pain/discomfort, blood tinged nasal mucus and nose bleed.
Percentage of Participants with Any Systemic Solicited Symptoms Anytime Post-Challenge | Up to 21 Days Post-Challenge
  Systemic signs or symptoms were defined as headache, fever, nausea, vomiting, abdominal cramps, diarrhea, malaise, and loss of appetite.
Percentage of Participants with Serious Adverse Events (SAEs) | 180 days following the last study vaccination (Up to Day 201)
  A SAE was any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Norwalk PAN-Ig Serum-ELISA Geometric Mean Titer (GMT) | Pre-Dose 1 and 21 Days Post Dose 1 and Dose 2
Norwalk PAN-Ig Serum-ELISA Geometric Mean Fold Rise (GMFR) | Pre-Dose 1 and 21 Days Post Dose 1 and Dose 2
  GMFR represents the geometric mean fold rise in antibody at post-dose compared to pre-dose 1.
Percentage of Participants with Norwalk PAN-Ig Serum-ELISA Seroresponse (4-Fold Rise) | Pre-dose 1 and 21 Days Post Dose 1 and 2
  4-Fold Rise represents the percentage of participants with at least a 4-Fold Rise in antibody at Day 21 post dose compared to pre-dose 1.
Norwalk IgG Serum-ELISA GMT | Pre-Dose 1 and 21 Days Post Dose 1 and Dose 2
Norwalk IgG Serum-ELISA GMFR | Pre-Dose 1 and 21 Days Post Dose 1 and Dose 2
  GMFR represents the geometric mean fold rise in antibody at post-dose compared to pre-dose 1.
Percentage of Participants with Norwalk IgG Serum-ELISA Seroresponse (4-Fold Rise) | Pre-Dose 1 and 21 Days Post Dose 1 and 2
  4-Fold Rise represents the percentage of participants with at least a 4-Fold Rise in antibody at Day 21 post dose compared to pre-dose 1.
Norwalk IgA Serum-ELISA GMT | Pre-Dose 1 and 21 Days Post Dose 1 and Dose 2
Norwalk IgA Serum-ELISA GMFR | Pre-Dose 1 and 21 Days Post Dose 1 and Dose 2
  GMFR represents the geometric mean fold rise in antibody at post-dose compared to pre-dose 1.
Percentage of Participants with Norwalk IgA Serum-ELISA Seroresponse | Pre-Dose 1 and 21 Days Post Dose 1 and 2
  4-Fold Rise represents the percentage of participants with at least a 4-Fold Rise in antibody at Day 21 post dose compared to pre-dose 1.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Atmar, MD, Principal Investigator — Baylor College of Medicine; David I Bernstein, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Clayton D Harro, MD, Principal Investigator — Johns Hopkins University; Mohamed S Al-Ibrahim, MD, Principal Investigator — SNBL Clinical Pharmacology Center, Inc.
Locations (3):
- United States (3):
  - SNBL, Baltimore, Maryland
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Atmar RL, Bernstein DI, Harro CD, Al-Ibrahim MS, Chen WH, Ferreira J, Estes MK, Graham DY, Opekun AR, Richardson C, Mendelman PM. Norovirus vaccine against experimental human Norwalk Virus illness. N Engl J Med. 2011 Dec 8;365(23):2178-87. doi: 10.1056/NEJMoa1101245. PMID 22150036